CLINICAL TRIAL: NCT04989868
Title: Effect of Trans-Nasal Afferent Loop Decompression on Post-Pancreaticoduodenectomy Pancreatic Fistula: An Open-label Randomized Controlled Trial
Brief Title: Effect of Trans-Nasal Afferent Loop Decompression on Post-Pancreaticoduodenectomy Pancreatic Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kuirong Jiang, Director of Pancreas Center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNALD
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Fistula; Pancreaticoduodenectomy; Complication of Surgical Procedure
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-Nasal Afferent Loop Decompression Arm (Experimental): Patients will receive trans-nasal afferent loop decompression after pancreaticoduodenectomy.
  Interventions: Procedure: Trans-Nasal Afferent Loop Decompression
- No Trans-Nasal Afferent Loop Decompression Arm (Active Comparator): Patients will NOT receive trans-nasal afferent loop decompression after pancreaticoduodenectomy.
  Interventions: Procedure: Without Trans-Nasal Afferent Loop Decompression

INTERVENTIONS:
Procedure: Trans-Nasal Afferent Loop Decompression — A 14Fr silicon tube with multiple side holes within the range of 15 cm from the tip will be placed into the afferent jejunal limb with its end close to the pancreaticojejunostomy (<3 cm) during the surgery. Continuous closed negative-pressure suction will be applied to that tube for 72 hours and after that the nasogastric tube will be removed. No nasogastric tube will be placed, or the nasogastric tube will be removed immediately after extubation.
  Arms: Trans-Nasal Afferent Loop Decompression Arm
Procedure: Without Trans-Nasal Afferent Loop Decompression — No decompression tube will be placed. No nasogastric tube will be placed, or the nasogastric tube will be removed immediately after extubation.
  Arms: No Trans-Nasal Afferent Loop Decompression Arm

SUMMARY:
Postoperative pancreatic fistula (POPF) is a major complication and an important cause of mortality after pancreaticoduodenectomy (PD). Trans-nasal afferent loop decompression technique (TNALD) may reduce the rate of POPF based on our previous retrospective study. The aim of this open-label randomized controlled trial is to determine whether TNALD is a protective factor against the development of POPF after PD.

DETAILED DESCRIPTION:
In our previous retrospective study, decompression of the afferent jejunal and pancreatic and biliary anastomoses with a special nasogastric tube and postoperative continuous closed negative pressure suction was shown to be associated with a reduction in overall POPF rate from 39% to 27% after PD. However, TNALD has the potential theoretical risk of increased morbidity including pulmonary complications and delayed gastric emptying.

The objective of this prospective randomized study is to evaluate the impact of trans-nasal afferent loop decompression on the incidence of complications after PD, especially POPF rate according to International Study Group of Pancreatic Surgery (ISGPS) 2016 updates. We hypothesize that the TNALD may prevent the development of POPF after PD. This study randomizes patients to TNALD versus no TNALD group. Subgroup analysis of the outcomes in different POPF risk groups is also planned.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for elective open pancreaticoduodenectomy with Child reconstruction
* Age > 18 years and ≤ 85 years
* Full agreement to participate and written informed consent is given

Exclusion Criteria:

* Emergent pancreaticoduodenectomy
* Laparoscopic pancreaticoduodenectomy or robotic pancreaticoduodenectomy, including transition to open approach
* Participant in other trials of pancreaticoduodenectomy with interfering interventions and/or endpoints
* Patient with severe co-morbidity(s) before surgery, including severe insufficiency in kidney, heart and/or liver, etc.
* Patient had medication history of corticosteroids over 3 days during last 30 days before surgery
* No need for pancreaticojejunostomy during pancreaticoduodenectomy (i.e. past left pancreatectomy, pancreaticogastrostomy, etc.), or pancreatic anastomosis cannot be reconstructed for any reason
* External stenting is used during the surgery for any reason
* Nasogastric tube is inserted and kept for postoperative gastric decompression
* In any situation that the placement of afferent loop decompression tube is medically inappropriate or not infeasible

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula (grade B+C) | up to 90 days after surgery
  Definition of postoperative pancreatic fistula was according ISGPS 2016 updates.

SECONDARY OUTCOMES:
Pancreatic fistula related complications | up to 90 days after surgery
  Including intra-abdominal infection and intra-abdominal fluid accumulation
Postoperative new-onset pulmonary complication | up to 14 days after surgery
  Including atelectasis, pleural effusion, pneumonitis
Other complications | up to 90 days after surgery
  Including postoperative hemorrhage, delayed gastric emptying, chyle leak, bile leak, sepsis, incision complication, deep vein thrombosis, pulmonary embolism, etc
Overall complication and severe complication | up to 90 days after surgery
  Overall complication (Clavien-Dindo ≥ grade I) and severe complication (Clavien-Dindo ≥ grade III)
Reintervention treatment | up to 90 days after surgery
  Number of patients with reintervention treatment for complications including percutaneous drainage, endoscopic procedure, angiographic procedure and reoperation
Mortality rate | up to 90 days after surgery
  Death for any reason
Length of postoperative stay | up to 90 days after surgery
  From surgery to discharge including ICU stay
Readmission | up to 90 days after surgery
  New admission within 90-days of discharge from hospital for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Jiang K Rong, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No